CLINICAL TRIAL: NCT05425849
Title: The Effect of Rose Oil Aromatherapy and Hand-Holding on Pain Due to Peripheral Intravenous Catheter Insertion: A Mixed Method Study
Brief Title: Pain Due to Peripheral Intravenous Catheter Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Tulay Basak, Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 394
Record Dates: First submitted 2022-06-11; First posted 2022-06-21 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): No attempt was made to reduce pain in the patients in the control group. Standard PIVC insertion procedure was applied.
- rose oil group (Experimental): After the patients in the rose aromatherapy group were placed in a sitting position, a face mask with 1-2 drops of rose oil was placed on the nose area. Then, the standard PIVC insertion procedure was applied. After the procedure, the patient's rose-scented mask was replaced with a standard mask.
  Interventions: Other: rose oil aromatherapy
- hand holding group (Experimental): After the patients in the hand-holding group were placed in a sitting position, the patient's family was asked to hold the patient's hand and not let it go until the procedure was over. Standard PIVC insertion procedure was applied.
  Interventions: Other: rose oil aromatherapy

INTERVENTIONS:
Other: rose oil aromatherapy — Aromatherapy refers to the medicinal or therapeutic use of essential oils absorbed through the skin or the olfactory system. The positive effects of social support, such as hand-holding, on anxiety and pain have been described
  Other Names: handholding
  Arms: hand holding group; rose oil group

SUMMARY:
This study aimed to evaluate the effectiveness of rose oil aromatherapy and hand-holding in reducing pain associated with peripheral intravenous catheters (PIVCs) insertion.

Study Hypothesis:

H0-1. The application of rose oil aromatherapy during the PIVC insertion procedure does not reduce the pain associated with the procedure.

H0-2. During the PIVC insertion procedure, the patient's family holding the patient's hand does not reduce the pain associated with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients voluntarily accepted to participate in the study,
* aged between 18-65,
* Turkish literate,
* PIVC placement planned,
* no hematoma, ecchymosis, scar and sensory change in the antecubital region,
* suitable for PIVC insertion with a 20 gauge (pink) catheter in the antecubital region,
* who did not take analgesic drugs for 24 hours and were accompanied by a member of the patient's family (spouse or child).
* patients with an Enhanced Adult DIVA (EA-DIVA) score below 8 for PIVC placement in a single intervention,
* the STAI score below 40

Exclusion Criteria:

* sensitive to smell and had problems in smelling,
* patients with epilepsy, asthma diagnosis,
* patients with a history of allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Pain Score | 1 minute-10 minutes
  Numeric Rating Scale was used. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Tulay Basak, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basak T, Demirtas A, Duman S. The effect of rose oil aromatherapy and hand-holding on pain due to peripheral intravenous catheter insertion. Explore (NY). 2024 Jan-Feb;20(1):62-69. doi: 10.1016/j.explore.2023.06.002. Epub 2023 Jun 7. PMID 37301653